CLINICAL TRIAL: NCT02173301
Title: A Phase 2, Randomized, Double-Blind, Multicenter, Parallel-Group, Placebo-Controlled Study to Assess the Efficacy and Safety of Three Dose Levels of XP23829 in Subjects With Moderate-to-Severe Chronic Plaque-Type Psoriasis
Brief Title: A Study to Assess the Efficacy and Safety of XP23829 in Subjects With Moderate-to-Severe Chronic Plaque-Type Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Collaborators: XenoPort, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XP-H-093
Record Dates: First submitted 2014-06-23; First posted 2014-06-24 (Estimated); Results first posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2017-11

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- XP23829 400 mg QD (once daily) (Experimental): After 4-week screening period, eligible subjects will be randomized to XP23829 400 mg QD for 12 weeks including titration period
  Interventions: Drug: XP23829 400 mg QD
- XP23829 800 mg QD (Experimental): After 4-week screening period, eligible subjects will be randomized to XP23829 800 mg QD for 12 weeks including titration period
  Interventions: Drug: XP 23829 800 mg QD
- XP23829 400 mg BID (twice daily) (Experimental): After 4-week screening period, eligible subjects will be randomized to XP23829 400 mg BID for 12 weeks including titration period
  Interventions: Drug: XP23829 400 mg BID
- Placebo (Placebo Comparator): After 4-week screening period, eligible subjects will be randomized to Placebo for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XP23829 400 mg QD — active dose 1
  Other Names: Tepilamide fumarate 400 mg QD; PPC-06 400 mg QD
  Arms: XP23829 400 mg QD (once daily)
Drug: XP 23829 800 mg QD — active dose 2
  Other Names: Tepilamide fumarate 800 mg QD; PPC-06 800 mg QD
  Arms: XP23829 800 mg QD
Drug: XP23829 400 mg BID — active dose 3
  Other Names: Tepilamide fumarate 400 mg BID; PPC-06 400 mg BID
  Arms: XP23829 400 mg BID (twice daily)
Drug: Placebo — control
  Arms: Placebo

SUMMARY:
The study objectives are the following:

1. To evaluate the efficacy of 3 doses of XP23829 compared to placebo for the treatment of moderate-to-severe chronic plaque-type psoriasis.
2. To evaluate the safety and tolerability of XP23829 in subjects with psoriasis.
3. To evaluate the pharmacodynamics (PD) of XP23829 through immunological analysis of peripheral blood samples.

DETAILED DESCRIPTION:
Study Design : This is a , multi-center, double blind, placebo-controlled, phase 2 (dose-finding) efficacy and safety study in which subjects with moderate-to- severe chronic plaque-type psoriasis will be randomized in a 1:1:1:1 allocation ratio to 1 of 3 active doses of XP23829 or placebo. Approximately 50 subjects will be enrolled into each treatment group.

Study Periods: The study includes a 4-week screening phase, a 12-week treatment phase (with 9 weeks of XP23829 or placebo at the maintenance dose), and a 4-week observational post-treatment follow-up phase. A treatment-free follow-up period is designed to evaluate safety and disease relapse and rebound.

Specifically, the study periods are as follows:

1. Screening Phase: Weeks -4 through 0
2. Treatment phase included:

   1. Titration Phase: Weeks 1 through 3
   2. Double-Blind Maintenance Phase: Weeks 4 through 12
3. Post-treatment follow-up: Weeks 13 through 16

Efficacy assessments will be performed in the clinic at Baseline (Visit 2) and at the end of Weeks 2, 4, 8, 12, 14, and 16.

Patient-reported outcome measures will be assessed in the clinic at Baseline and at Week 12.

Blood samples for pharmacodynamic (PD) assessments will be collected at Baseline and at Weeks 4, 8, 12 and 16. PD assessments will be conducted in all subjects, with the intent of evaluating psoriasis-associated inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, age ≥ 18.
2. Stable, moderate-to-severe plaque-type psoriasis diagnosed for at least 6 months prior to randomization (no morphology changes or significant flares of disease activity in the last 6 months in the opinion of the investigator).
3. Severity of disease meeting all of the following three criteria prior to randomization:

   1. Psoriasis Area and Severity Index (PASI) score of 12 or greater
   2. Total Body Surface Area (BSA) affected by plaque psoriasis of 10% or greater
   3. Static Physician's Global Assessment (sPGA) score of 3 or greater
4. Must be a candidate for phototherapy and/or systemic therapy for psoriasis.

Exclusion Criteria:

1. Subjects with current inverse, erythrodermic, predominantly guttate, or pustular psoriasis.
2. Subjects with current drug-induced or drug-exacerbated psoriasis.
3. Subjects with moderate-to-severe psoriatic arthritis of any type; and subjects with mild psoriatic arthritis, who require systemic disease-modifying therapy.
4. Subjects with unstable or significant illness, including the presence of laboratory abnormalities at screening that in the opinion of the investigator would place the subject at unacceptable risk if he/she were to participate in the study.
5. Any skin condition (e.g. eczema) which confounds the ability to interpret data from the study.
6. Treatment with a topical anti-psoriatic therapy within 14 days prior to randomization (including topical steroids, topical vitamin A or D analog preparations, tacrolimus, pimecrolimus, or anthralin).
7. Phototherapy or prolonged sun exposure or use of ultraviolet (UV) light sources within 28 days of randomization.
8. Use of investigational or approved biologic treatments that are known to affect psoriasis, such as adalimumab, etanercept, golimumab or infliximab within 12 weeks of randomization and ustekinumab within 24 weeks of randomization.
9. Use of systemic medications (non-biologics) that are known to affect psoriasis (including but not limited to oral corticosteroids, cyclosporine, methotrexate, lithium, and beta-adrenergic blockers) within 4 weeks of randomization, or 5 half-lives, whichever is longer.
10. Prior treatment with Dimethyl Fumarate (Fumaderm® or Tecfidera®) or any other Fumaric Acid Ester (FAE) containing products.
11. Have failed (due to inadequate response) more than 3 approved systemic agents for the treatment of psoriasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dmitri Lissin, M.D., Study Director — XenoPort, Inc.
Locations (28):
- United States (28):
  - XenoPort Investigational Site, Birmingham, Alabama
  - XenoPort Investigational Site, Phoenix, Arizona
  - XenoPort Investigational Site, Hot Springs, Arkansas
  - XenoPort Investigational Site, Encinitas, California
  - XenoPort Investigational Site, Fremont, California
  - XenoPort Investigational Site, Fullerton, California
  - XenoPort Investigational Site, Denver, Colorado
  - XenoPort Investigational Site, Snellville, Georgia
  - XenoPort Investigational Site, Buffalo Grove, Illinois
  - XenoPort Investigational Site, Carmel, Indiana
  - XenoPort Investigational Site, South Bend, Indiana
  - XenoPort Investigational Site, Overland Park, Kansas
  - XenoPort Investigational Site, Louisville, Kentucky
  - XenoPort Investigational Site, Owensboro, Kentucky
  - XenoPort Investigational Site, Boston, Massachusetts
  - XenoPort Investigational Site, Watertown, Massachusetts
  - XenoPort Investigational Site, Troy, Michigan
  - XenoPort Investigational Site, Warren, Michigan
  - XenoPort Investigational Site, Omaha, Nebraska
  - XenoPort Investigational Site, East Windsor, New Jersey
  - XenoPort Investigational Site, Verona, New Jersey
  - XenoPort Investigational Site, Rochester, New York
  - XenoPort Investigational Site, Stony Brook, New York
  - XenoPort Investigational Site, High Point, North Carolina
  - XenoPort Investigational Site, Goodlettsville, Tennessee
  - XenoPort Investigational Site, Dallas, Texas
  - XenoPort Investigational Site, San Antonio, Texas
  - XenoPort Investigational Site, West Jordan, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- XP23829 800 mg QD (Once Daily): After 4-week screening period, eligible subjects will be randomized to XP23829 800 mg QD for 12 weeks including titration period
  XP 23829 800 mg QD: active dose 2
Period: Overall Study
Arm/Group | XP23829 400 mg QD (Once Daily) | XP23829 800 mg QD (Once Daily) | XP23829 400 mg BID (Twice Daily) | Placebo
Started | 49 | 55 | 48 | 48
Completed | 29 | 32 | 28 | 33
Not Completed | 20 | 23 | 20 | 15
Not completed — Adverse Event | 7 | 8 | 13 | 5
Not completed — Withdrawal by Subject | 8 | 10 | 4 | 8
Not completed — Lost to Follow-up | 4 | 4 | 2 | 2
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Subject unable to return for week 16 assessment within Sponsor timelines for study completion | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | XP23829 400 mg QD (Once Daily) | XP23829 800 mg QD (Once Daily) | XP23829 400 mg BID (Twice Daily) | Placebo | Total
Number analyzed (Participants) | 49 | 55 | 48 | 48 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (11.89) | 47.7 (10.55) | 51.8 (13.80) | 51.1 (13.66) | 50.3 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 23 | 16 | 14 | 70
  Male | 32 | 32 | 32 | 34 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 11 | 1 | 31
  Not Hispanic or Latino | 37 | 48 | 37 | 47 | 169
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 1 | 3
  Asian | 0 | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 3 | 1 | 2 | 10
  White | 44 | 48 | 45 | 44 | 181
  More than one race | 1 | 1 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline PASI score [Mean (Standard Deviation); unit: units on a scale] — The PASI is a measure of the average redness, thickness, and scaliness of the lesions (each graded on a 0-4 scale) and is weighted by the area of involvement. The minimum possible score on this scale is '0', while the maximum score on this scale is 72. A lower score on this scale at the end of the study indicates an improvement in the condition of subject.
  PASI score assessed at Baseline Visit
  units on a scale | 18.32 (7.413) | 18.19 (7.977) | 17.51 (4.791) | 19.13 (7.671) | 18.28 (7.082)
Baseline sPGA [Count of Participants; unit: Participants] — Score Grade : Definition - 0 Clear: No signs of psoriasis Almost clear: No thickening to minimal plaque elevation; Normal to slight pink coloration/faint erythema; Focal to minimal scaling Mild: Slight elevation/thickening; Pink to light red coloration; Predominantly fine scaling partially or mostly covering lesions Moderate: Clearly distinguishable/distinct thickening; Definite red coloration; Coarse scaling covering most plaques Severe: Marked thickening with hard/sharp edges; Bright to deep dark red coloration; Thick/coarse scaling covering almost all or all lesions
  sPGA atbaseline
  Participants
    3 Moderate | 32 | 39 | 34 | 34 | 139
    4 Severe | 17 | 16 | 14 | 14 | 61
Baseline Body Surface Area involved [Mean (Standard Deviation); unit: percentage] — Percentage of the subject's total body surface area (BSA) that is involved by lesions of plaque psoriasis .
  Percentage of total BSA involved by psoriasis lesions at Baseline
  percentage | 22.90 (13.324) | 23.79 (15.283) | 23.08 (14.585) | 26.44 (16.260) | 24.04 (14.860)
Has Used Systemic Biologics? [Count of Participants; unit: Participants] — Subjects who have used one or more systemic biologic treatment(s) for their plaque psoriasis in the past.
  This information is collected at Screening/ Baseline Visit
  Participants
    No | 32 | 34 | 30 | 35 | 131
    Yes | 17 | 21 | 18 | 13 | 69
Body Weight [Mean (Standard Deviation); unit: kilograms] — Subject's body weight as of Baseline Visit
  kilograms | 95.22 (25.710) | 101.68 (26.142) | 101.08 (27.207) | 97.08 (25.136) | 98.85 (26.007)

OUTCOME MEASURES:

1. Primary Outcome: • The Percent Change in PASI (Psoriasis Area and Severity Index) Score From Baseline
Description: The PASI is a measure of the average redness, thickness, and scaliness of the lesions (each graded on a 0-4 scale) and is weighted by the area of involvement. The minimum possible score on this scale is '0', while the maximum score on this scale is 72. A lower score on this scale at the end of the study indicates an improvement in the condition of subject.
Time Frame: 12 Weeks
Population: modified Intent-to-Treat population Observed cases analysis
Measure: Least Squares Mean (Standard Error); unit: percentage change from baseline
Arm/Group | XP23829 400 mg QD (Once Daily) | XP23829 800 mg QD (Once Daily) | XP23829 400 mg BID (Twice Daily) | Placebo
Number analyzed (Participants) | 48 | 53 | 46 | 47
percentage change from baseline | -38.1 (5.07) | -48.2 (5.06) | -50.7 (5.50) | -25.0 (5.06)
Statistical Analysis 1: Comparison: XP23829 400 mg QD (Once Daily) vs Placebo; Test type: Superiority; p = 0.066, Mixed Models Analysis; Restricted Maximum Likelihood (REML) - an REML-based mixed model for repeated measures (MMRM) with and with baseline PASI score as covariate
Statistical Analysis 2: Comparison: XP23829 800 mg QD (Once Daily) vs Placebo; Test type: Superiority; p = 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: XP23829 400 mg BID (Twice Daily) vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: • Proportion of Subjects Who Achieve a Reduction of 75% or Greater From Baseline in PASI (PASI-75)
Description: The percentage of subjects who achieve a reduction of 75% or greater from Baseline in the Psoriasis Area and Severity Index score (PASI-75) at efficacy assessments conducted at Weeks 2, 4, 8, 12, 14 and 16. The PASI is a measure of the average redness, thickness, and scaliness of the lesions (each graded on a 0-4 scale) and is weighted by the area of involvement. The minimum possible score on this scale is '0', while the maximum score on this scale is 72. A lower score on this scale at the end of the study indicates an improvement in the condition of subject.
Time Frame: Weeks 2, 4, 8, 12, 14 and 16
Population: modified Intent-to-treat population with last observation carried forward imputation for missing values
Measure: Count of Participants; unit: Participants
Arm/Group | XP23829 400 mg QD (Once Daily) | XP23829 800 mg QD (Once Daily) | XP23829 400 mg BID (Twice Daily) | Placebo
Number analyzed (Participants) | 48 | 53 | 46 | 47
Participants
  Week 2: number analyzed (Participants) | 46 | 50 | 46 | 43
  Week 2 | 1 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 47 | 50 | 46 | 44
  Week 4 | 2 | 0 | 2 | 0
  Week 8: number analyzed (Participants) | 47 | 50 | 46 | 44
  Week 8 | 3 | 2 | 5 | 2
  Week 12: number analyzed (Participants) | 47 | 50 | 46 | 44
  Week 12 | 6 | 7 | 10 | 4
  Week 14 | 6 | 4 | 6 | 3
  Week 16 | 3 | 3 | 6 | 2
Statistical Analysis 1: Comparison: XP23829 400 mg QD (Once Daily) vs Placebo; Week 12 comparison; Test type: Superiority; p = 0.501, Regression, Logistic
Statistical Analysis 2: Comparison: XP23829 800 mg QD (Once Daily) vs Placebo; Week 12 comparison; Test type: Superiority; p = 0.340, Regression, Logistic
Statistical Analysis 3: Comparison: XP23829 400 mg BID (Twice Daily) vs Placebo; Week 12 comparison; Test type: Superiority; p = 0.075, Regression, Logistic

3. Secondary Outcome: • Proportion of Subjects Who Achieve a sPGA (Static Physician's Global Assessment) Score of Clear or Almost Clear
Description: The Percentage of subjects who achieve the static Physician's Global Assessment (sPGA) score of 'clear' or 'almost clear' (sPGA score 0 or 1) at efficacy assessments conducted at Weeks 2, 4, 8, 12, 14 and 16.
  Score Grade : Definition - 0 Clear: No signs of psoriasis
  1. Almost clear: No thickening to minimal plaque elevation; Normal to slight pink coloration/faint erythema; Focal to minimal scaling
  2. Mild: Slight elevation/thickening; Pink to light red coloration; Predominantly fine scaling partially or mostly covering lesions
  3. Moderate: Clearly distinguishable/distinct thickening; Definite red coloration; Coarse scaling covering most plaques
  4. Severe: Marked thickening with hard/sharp edges; Bright to deep dark red coloration; Thick/coarse scaling covering almost all or all lesions
  A lower score on this scale at the end of the study indicates an improvement in the disease condition.
Time Frame: Weeks 2, 4, 8, 12, 14 and 16
Population: modified 'Intent-to-treat' population using Last Observation Carried Forward method to impute missing observations
Measure: Count of Participants; unit: Participants
Arm/Group | XP23829 400 mg QD (Once Daily) | XP23829 800 mg QD (Once Daily) | XP23829 400 mg BID (Twice Daily) | Placebo
Number analyzed (Participants) | 48 | 53 | 46 | 47
Participants
  Week 2: number analyzed (Participants) | 46 | 50 | 46 | 43
  Week 2 | 0 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 47 | 50 | 46 | 44
  Week 4 | 1 | 1 | 0 | 0
  Week 8: number analyzed (Participants) | 47 | 50 | 46 | 44
  Week 8 | 2 | 2 | 1 | 2
  Week 12: number analyzed (Participants) | 47 | 50 | 46 | 44
  Week 12 | 5 | 3 | 3 | 2
  Week 14 | 5 | 2 | 3 | 1
  Week 16 | 5 | 1 | 4 | 1
Statistical Analysis 1: Comparison: XP23829 400 mg QD (Once Daily) vs Placebo; Week 12 comparison; Test type: Superiority; p = 0.229, Regression, Logistic
Statistical Analysis 2: Comparison: XP23829 800 mg QD (Once Daily) vs Placebo; Week 12 comparison; Test type: Superiority; p = 0.604, Regression, Logistic
Statistical Analysis 3: Comparison: XP23829 400 mg BID (Twice Daily) vs Placebo; Week 12 comparison; Test type: Superiority; p = 0.573, Regression, Logistic

ADVERSE EVENTS:
Time Frame: Baseline to Week 16 or study discontinuation
Description: Adverse Events are reported in the safety population ( which is identical to the randomized subject and intent-to treat populations)
Arm/Group | XP23829 400 mg QD (Once Daily) | XP23829 800 mg QD (Once Daily) | XP23829 400 mg BID (Twice Daily) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/55 | 0/48 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/49 | 1/55 | 1/48 | 0/48
Other Adverse Events (participants affected / at risk) | 36/49 | 42/55 | 37/48 | 29/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XP23829 400 mg QD (Once Daily) (N=49) | XP23829 800 mg QD (Once Daily) (N=55) | XP23829 400 mg BID (Twice Daily) (N=48) | Placebo (N=48)
Abdominal Adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | NA (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XP23829 400 mg QD (Once Daily) (N=49) | XP23829 800 mg QD (Once Daily) (N=55) | XP23829 400 mg BID (Twice Daily) (N=48) | Placebo (N=48)
Diarrhea (Gastrointestinal disorders) | 11 | 22 | 19 | 7
Nausea (Gastrointestinal disorders) | 6 | 4 | 10 | 6
Abdominal pain (Gastrointestinal disorders) | 1 | 7 | 11 | 2
Flushing (Vascular disorders) | 4 | 3 | 2 | 3
Headache (Nervous system disorders) | 2 | 3 | 5 | 2
Vomiting (Gastrointestinal disorders) | 3 | 7 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 3 | 2
Flatulence (Gastrointestinal disorders) | 2 | 5 | 3 | 0
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 4 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 4 | 2 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 3 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication would have to be collaborative effort between Sponsor and Investigators